CLINICAL TRIAL: NCT02300857
Title: Effects of Macronutrient Diet Composition on Brain Reward Activity
Brief Title: Effects of Macronutrient Diet on Brain Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Boston Children's Hospital (Other); Nutrition Science Initiative (Other); New Balance Foundation (Other); Boston Medical Center (Other); Framingham State University (Other)
Responsible Party: Principal Investigator, Laura M. Holsen, Assistant Professor of Psychiatry, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2014P001880
Record Dates: First submitted 2014-11-20; First posted 2014-11-25 (Estimated); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Diet, Carbohydrate-Restricted; Diet, High-Protein Low-Carbohydrate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low carbohydrate diet (Active Comparator)
  Interventions: Behavioral: Low carbohydrate diet
- Moderate carbohydrate diet (Active Comparator)
  Interventions: Behavioral: Moderate carbohydrate diet
- High carbohydrate diet (Active Comparator)
  Interventions: Behavioral: High carbohydrate diet

INTERVENTIONS:
Behavioral: Low carbohydrate diet — Feeding study. Composition (by proportion of calories): 20% carbohydrate, 60% fat, 20% protein
  Arms: Low carbohydrate diet
Behavioral: Moderate carbohydrate diet — Feeding study. Composition (by proportion of calories): 40% carbohydrate, 40% fat, 20% protein
  Arms: Moderate carbohydrate diet
Behavioral: High carbohydrate diet — Feeding study. Composition (by proportion of calories): 60% carbohydrate, 20% fat, 20% protein
  Arms: High carbohydrate diet

SUMMARY:
This study will evaluate the effect of macronutrient diets on brain activity in homeostatic and mesolimbic reward regions.

DETAILED DESCRIPTION:
A question critical to the field of obesity is "what causes overweight and obese individuals to overeat?" One common explanation holds that weight gain at the population-level is caused by increases in the widespread availability of highly palatable foods. An alternative explanation is that the biological effects of the modern diet produce effects in the central nervous system and periphery that augment homeostatic and hedonic hunger. Reducing glycemic load preferentially maintains total energy expenditure during weight-loss maintenance (Ebbeling et al., 2012), and this group of investigators previously showed that in the late postprandial period, a nutrient-controlled high glycemic load vs. low glycemic load meal increases resting regional cerebral blood flow in the nucleus accumbens (Lennerz et al., 2013), part of the mesoaccumbal reward circuitry implicated in craving and addiction. However, the effects of macronutrient composition on blood flow to and activity in homeostatic and reward-related brain regions cannot be fully ascertained from studies of acute ingestion of a single macronutrient, because these do not generalize to mixed-nutrient meals consumed as part of typical American diets. Further, retrospective designs that rely on participant report of frequency of recent macronutrient ingestion and prospective designs with limited duration of diet prescription cannot address the critical question of the long-term, cumulative effects of dietary composition on brain function. Therefore, the investigators propose an approach to identifying brain responses to randomized, mixed-meal diets of varying macronutrient composition during long-term weight-loss maintenance on these diets, using arterial spin labeling (ASL) for regional cerebral blood flow (rCBF) and blood-oxygen-level-dependent (BOLD)-based functional connectivity.

To explore these outcomes, the investigators will partner with the ongoing Framingham State Food Study (NCT02068885): Following weight loss on a standard diet, 150 overweight or obese adults (aged 18 to 65 years) will be randomized to one of three weight-loss maintenance diets varying in carbohydrate to fat ratios for 20 weeks. Investigators will invite subjects already enrolled in the Framingham State Food Study to participate with a goal of enrolling 75 subjects (aiming to be equally divided per diet group following randomization to assigned test diet in the parent study). Participants will complete 1 morning visit to the MRI imaging center at Brigham and Women's Hospital approximately 14-20 weeks into the weight maintenance test diet phase. During the visit, they will undergo a fasting baseline brain imaging session, consume their assigned diet breakfast meal, and undergo a late postprandial brain imaging session. Participants will additionally provide frequent ratings of their food cravings, mood, and anxiety level throughout the visit. The main outcomes will be resting blood flow to the nucleus accumbens and connected striatal regions in the late postprandial period, with additional secondary and other outcomes including blood flow to the hypothalamus and connectivity between the hypothalamus during the late postprandial period.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 55 years
* BMI ≥ 23 kg/m2
* BMI < 45 kg/m2 and weight ≤ 300 lbs (136 kg)
* Medical clearance from a primary care provider
* Student or employee at Framingham State University throughout enrollment in the study
* Community-based participants from the greater Framingham and Assabet Valley communities
* Willing and able to eat and drink only the foods and beverages on the study menus
* Willing to eat in the dining hall
* Willing to abstain from consuming alcohol during participation

Additional Inclusion Criteria:

* Body circumference of <64 in
* Willingness to undergo 2, 30-minute MRI scans

Exclusion Criteria (as detailed in Framingham State Food Study, NCT02068885):

* Change in body weight exceeding ±10% during prior year
* Recent adherence to a special diet
* Recent adherence to a vigorous physical activity regimen (e.g., participation in a varsity sport)
* Chronic use of any medication or dietary supplement that could affect study outcomes
* Current smoking (1 cigarette in the last week)
* Heavy baseline alcohol consumption or history of binge drinking
* Physician diagnosis of a major medical/psychiatric illness or eating disorder
* Abnormal blood glucose, TSH, CBC, BUN, Creatinine
* ALT greater than 150% of the normal upper limit
* Plans for a vacation during the study that would preclude adherence to prescribed diet
* Additional exclusions for female participants: Irregular menstrual cycles; any change in birth control medication during the 3 months prior to enrollment; pregnancy or lactation during the 12 months prior to enrollment

Additional Exclusion Criteria:

* Previous bariatric surgery
* Other contraindications to MRI scanning (severe claustrophobia/extensive orthopedic hardware/pacemaker, cerebral aneurysm clip)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Blood flow to the nucleus accumbens and connected striatal regions | 14-20 weeks after initiation of test diet
  Regional cerebral blood flow (rCBF) measured using arterial spin labeling (ASL) at rest, in neuroanatomically-defined a priori regions (nucleus accumbens, caudate, putamen).

SECONDARY OUTCOMES:
Blood flow to the hypothalamus | 14-20 weeks after initiation of test diet
  Regional cerebral blood flow (rCBF) measured using arterial spin labeling (ASL) at rest, in neuroanatomically-defined a priori regions (hypothalamus).
Functional connectivity between the hypothalamus and nucleus accumbens | 14-20 weeks after initiation of test diet
  Blood-oxygen-level-dependent (BOLD) fMRI connectivity between neuroanatomically-defined regions of interest (hypothalamus, nucleus accumbens), measured during rest.

CONTACTS AND LOCATIONS:
Overall Officials: Laura M. Holsen, Ph.D., Principal Investigator — Brigham and Women's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lennerz BS, Alsop DC, Holsen LM, Stern E, Rojas R, Ebbeling CB, Goldstein JM, Ludwig DS. Effects of dietary glycemic index on brain regions related to reward and craving in men. Am J Clin Nutr. 2013 Sep;98(3):641-7. doi: 10.3945/ajcn.113.064113. Epub 2013 Jun 26. PMID 23803881
- [Derived] Holsen LM, Hoge WS, Lennerz BS, Cerit H, Hye T, Moondra P, Goldstein JM, Ebbeling CB, Ludwig DS. Diets Varying in Carbohydrate Content Differentially Alter Brain Activity in Homeostatic and Reward Regions in Adults. J Nutr. 2021 Aug 7;151(8):2465-2476. doi: 10.1093/jn/nxab090. PMID 33852013
- See also: Link to the Framingham State Food Study (parent study) — http://clinicaltrials.gov/show/NCT02068885